CLINICAL TRIAL: NCT02672228
Title: Feasibility of the Vapor Nanobubble Technology (MalariSense) for Malaria Diagnostics
Brief Title: Feasibility of the Vapor Nanobubble Technology for Malaria Diagnostics (MalariaSense)
Acronym: MalariaSense
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Precision Acoustics ltd UK (Unknown); Standa, UAB Lithuania (Unknown); X Instruments LLC, CA, USA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCC 1430
Record Dates: First submitted 2015-09-14; First posted 2016-02-03 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MalariaSense device (Experimental): This study will involve the evaluation of a medical diagnostic device. All participants enrolled in the study will be assessed for malaria using MalariSense Technology and will aslo get rapid diagnostic tests (RDTs), microscopy, PCR
  Interventions: Device: MalariaSense device

INTERVENTIONS:
Device: MalariaSense device — All participants enrolled in the study will be assessed for malaria using the intervention device called MalariaSense technology

SUMMARY:
This is a proof of concept study that will evaluate the feasibility of a vapor nanobubble technology (MalariSense) for malaria diagnostics. The MalariSense technology will use a highly innovative approach based on the transdermal non-invasive detection of vapor nanobubbles produced by the excitation of malaria-specific hemozoin by safe, low-energy laser pulse. The objectives of this study will be to determine the sensitivity and specificity of MalariSense in diagnosing malaria in malaria suspected cases attending a health facility in The Gambia and to identify factors influencing the diagnostic accuracy of MalariSense

DETAILED DESCRIPTION:
This is a proof of concept study that will evaluate the feasibility of a vapor nanobubble technology (MalariSense) for malaria diagnostics. The primary objective is to determine the sensitivity of MalariSense against microscopy in diagnosing malaria in malaria suspected cases attending a health facility in The Gambia. The secondary objectives include the following;

1. To determine the sensitivity of MalariSense against PCR in diagnosing malaria in malaria suspected cases attending a health facility in The Gambia
2. To determine the specificity of MalariSense in diagnosing malaria in malaria suspected cases attending a health facility in The Gambia.
3. To identify factors influencing the diagnostic accuracy of MalariSense
4. To validate the protocol for a blood vessel identification for the test and assess the safety of the prototype The study site will be Basse in the Eastern region of The Gambia. The study will be conducted during the malaria transmission season (August to December 2015). Participants will be patients with suspected uncomplicated malaria presenting to the outpatient department of Basse Health centre. At baseline, suspected malaria cases (clinical assessment) will be asked to provide informed consent and then transferred to the MRC Basse field station where a finger prick blood sample will be collected for a malaria rapid diagnostic test (RDT), microscopy and on filter paper for subsequent molecular studies. In addition, they will be tested using the Malarisense Technology. Measurements will be taken from the wrist, ear lobe and finger tips. The laboratory prototype of the device will include three major components: pulsed laser with the fiber output, integrated handheld probe with the fiber launch in the center and an ultrasound sensor with pre-amplifier, and the signal acquisition hardware with software.

The study will enrol a total sample size of 50 patients with confirmed malaria. It is estimated that about 125 to 167 suspected cases will need to be screened/tested to get this sample size. The Sample size will be increased by 10% to allow for any missing values - therefore up to 185 suspected cases screened. In addition, a convenience sample of 30 malaria negative participants will be enrolled for comparisons between malaria positive and malaria negative populations. RDT positive patients will be provided with antimalarial treatment while the others will receive treatment according to their condition. Microscopy and species-specific PCR will be performed later. Microscopy results will be taken as the gold standard.

There will not be any active follow up. Study participants will be asked to come back 2 days after the test, or earlier if they notice a problem.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the health facility with suspected uncomplicated malaria
* Provision of informed consent

Exclusion Criteria:

* Neonates and under 12 months old
* Pregnant women

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
"Hemozoin-generated vapour nanobubble (H-VNB) amplitude thresholds among malaria infected and uninfected individuals" | Day 1

SECONDARY OUTCOMES:
Safety profile of Malarisense technology for malaria diagnosis | Day 1 - Day 3
  Safety of the MalariSense Technology for malaria diagnosis over 3 days of observation
Correlation of incidence rate ratio of hemozoin-positive traces with level of parasite density as determined by microscopy | Day1 - Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Umberto D'alessandro, PhD, MD, Principal Investigator — Medical Research Council Unit, The Gambia
Locations (1):
- Basse Health Centre, Basse, Upper River Region, The Gambia